CLINICAL TRIAL: NCT07085208
Title: Derivation and Verification of Hemodynamic Clinical Subphenotypes in Patients Undergoing Cardiac Surgery Under Unsupervised Machine Learning
Brief Title: Derivation and Validation of Hemodynamic Phenotypes of Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20250224-KS-04
Record Dates: First submitted 2025-07-15; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-02

CONDITIONS: Phenotyping; Machine Learning; Cardiac Surgery; Hemodynamic Parameters
MeSH Terms: interventions — Unsupervised Machine Learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Unsupervised Machine Learning for Clinical Phenotyping — This is a data-driven study that uses an unsupervised machine learning algorithm to perform clustering on patient multimodal features. These features include: preoperative demographics, comorbidities, and laboratory data; surgical information; and high-resolution intraoperative data, most notably continuous vital sign trajectories.

SUMMARY:
Background & Objective:

Cardiac surgery patients differ significantly in their health conditions and how they react during operations. Standard risk assessments before surgery often miss the real-time changes happening inside a patient's body during the procedure, which can affect their recovery. Therefore, researchers conducted this study to find different groups (phenotypes) of patients who face varying risks for poor outcomes. They did this by using advanced computer learning techniques to analyze a lot of detailed health information collected both before and during surgery.

Methods:

This was a study that looked back at patient records from several hospitals. Researchers gathered a large amount of patient information from before surgery, including their basic health details and lab results. They also collected very detailed measurements of patients' vital signs taken during surgery, noting how these changed over time. Then, a computer program that can find patterns without being told what to look for (unsupervised hierarchical clustering) was used to sort patients into distinct groups based on this combined data.

Clinical Relevance:

This study expects to show that using data to identify patient groups can reveal differences that traditional methods miss. These new patient groups, which are based on how their blood flow and vital signs behave, offer a new way to understand risks in real-time. This could help doctors to predict problems more accurately and create personalized care plans for each patient around the time of surgery, which has great potential for practical use in hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients who underwent cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Incomplete information on surgical procedures,
* With History of prior cardiac surgery or underwent second surgery during the same hospitalization
* Insufficient valid perioperative vital sign monitoring data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 years or older who underwent cardiac surgery with CPB were identified from each database.
Sampling Method: Non-Probability Sample
Enrollment: 10847 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Acute organ dysfunction | Within 7 days post-surgery for acute liver failure and acute kidney inkury, and 90 days for postoperative acute kidney disease
  including postoparative acute liver failure and acute kidney injury (up to 7 days postoperative), and acute kidney disease(up to 90 days postoperative)

SECONDARY OUTCOMES:
Total LOS and ICU-LOS | up to 90 days post-surgery
  Length of hospital stay and length of ICU stay
In-hospital mortality | up to 90 days postoperative, from the end of surgery until patient discharge
  All-cause in-hospital mortality